CLINICAL TRIAL: NCT05039489
Title: A Study on the Brain Mechanism of cTBS in Improving Medication-resistant Auditory Hallucinations in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Guo Wenbin, Professor of Psychiatry Department of Psychiatry of the Second Xiangya Hospital, Central South University, Central South University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 82171508
Record Dates: First submitted 2021-08-31; First posted 2021-09-09 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Schizophrenia
Keywords: Medication-Resistant Auditory Hallucinations; Continuous theta burst stimulation，cTBS; Neuroimaging
MeSH Terms: conditions — Schizophrenia | interventions — Antipsychotic Agents; Magnetic Resonance Spectroscopy; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- The schizophrenia patients with medication-resistant auditory hallucinations (Experimental): Drug + cTBS intervention (the left cerebellum Crus II as the stimulation target)
  Interventions: Drug: Antipsychotic drugs; Device: cTBS （the left cerebellum Crus II as the stimulation target）
- The schizophrenia patients with general auditory hallucinations (Active Comparator): Drug intervention
  Interventions: Drug: Antipsychotic drugs
- The healthy controls (No Intervention): MRI scan at baseline and no drugs treatment
- Drug + cTBS intervention: the first-episode schizophrenia patients with auditory hallucinations (Experimental): Drug + cTBS intervention (the left temporoparietal cortex as the stimulation target)
  Interventions: Drug: Antipsychotic drugs; Device: cTBS（the left temporoparietal cortex as the stimulation target）
- Drug intervention: the first-episode schizophrenia patients with auditory hallucinations (Active Comparator): Drug intervention
  Interventions: Drug: Antipsychotic drugs
- The schizophrenia patients with medication-resistant auditory hallucinations from the fourth arm (Experimental): Drug + cTBS intervention (the left cerebellum Crus II as the stimulation target)
  Interventions: Drug: Antipsychotic drugs; Device: cTBS （the left cerebellum Crus II as the stimulation target）

INTERVENTIONS:
Drug: Antipsychotic drugs — Stable antipsychotic medication 4 weeks before and during the treatment. Chlorpromazine (CPZ) equivalent dosages were calculated for second- and first-generation antipsychotic drugs
  Other Names: MRI scan
  Arms: Drug + cTBS intervention: the first-episode schizophrenia patients with auditory hallucinations; Drug intervention: the first-episode schizophrenia patients with auditory hallucinations; The schizophrenia patients with general auditory hallucinations; The schizophrenia patients with medication-resistant auditory hallucinations; The schizophrenia patients with medication-resistant auditory hallucinations from the fourth arm
Device: cTBS（the left temporoparietal cortex as the stimulation target） — Participants received 3 daily sessions of cTBS treatment. One session of cTBS was 40 seconds in duration and consisted of 3-pulse bursts at 50 Hz repeated every 200 milliseconds (5 Hz) until a total of 600 pulses was reached. To achieve cumulative aftereffects, this protocol was repeated 3 times and (1800 pulses in total) separated by two 15 minute breaks
  Other Names: MRI scan
  Arms: Drug + cTBS intervention: the first-episode schizophrenia patients with auditory hallucinations
Device: cTBS （the left cerebellum Crus II as the stimulation target） — Participants received 3 daily sessions of cTBS treatment. One session of cTBS was 40 seconds in duration and consisted of 3-pulse bursts at 50 Hz repeated every 200 milliseconds (5 Hz) until a total of 600 pulses was reached. To achieve cumulative aftereffects, this protocol was repeated 3 times and (1800 pulses in total) separated by two 15 minute breaks
  Other Names: MRI scan
  Arms: The schizophrenia patients with medication-resistant auditory hallucinations; The schizophrenia patients with medication-resistant auditory hallucinations from the fourth arm

SUMMARY:
This study is dedicated to exploring the brain mechanism of medication-resistant auditory hallucinations and developing effective treatment methods for them by using both cross-sectional and longitudinal designs. The continuous theta burst stimulation(cTBS) treatment mode, with the left cerebellum Crus II as the stimulation target, is applied to treat the schizophrenia patients with the medication-resistant auditory hallucinations. At the same time, the first-episode schizophrenia patients with auditory hallucinations were recruited as a test cohort to examine that brain mechanism of general auditory hallucinations in schizophrenia may be the structural and functional abnormalities in the temporoparietal circuit.

DETAILED DESCRIPTION:
Previous studies have shown that repetitive transcranial magnetic stimulation (rTMS) targeted at the temporal-parietal junction can effectively treat genenal auditory hallucinations in schizophrenia, but it is not the case for medication-resistant auditory hallucinations. Studies suggested that rTMS targeted at the left Crus II might be effective for medication-resistant auditory hallucinations. This study is dedicated to exploring the brain mechanism of medication-resistant auditory hallucinations and developing effective treatment methods for them by using both cross-sectional and longitudinal designs. The continuous theta burst stimulation(cTBS) treatment mode, with the left cerebellum Crus II as the stimulation target, is applied to treat the schizophrenia patients with the medication-resistant auditory hallucinations. Assessment with symptomatology, neuropsychology, neuroimaging, and machine learning methods is utilized to examine the investigators hypothesis that structural and functional abnormalities of the cerebral cortico-cerebellar-thalamic-cortical circuit (CCTCC) may contribute to brain mechanism of medication-resistant auditory hallucinations in schizophrenia. At the same time, the first-episode schizophrenia patients with auditory hallucinations were recruited as a test cohort to examine that brain mechanism of general auditory hallucinations in schizophrenia may be the structural and functional abnormalities in the temporoparietal circuit, whereas structural and functional abnormalities of the CCTCC may contribute to brain mechanism of medication-resistant auditory hallucinations in schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. 18-45 years old, right-handed
3. Meet the diagnostic criteria for schizophrenia according to the Structural Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V)
4. After a sufficient course of antipsychotic treatment (more than 6 weeks, two or more antipsychotic drugs, at least one of which is the second generation of atypical antipsychotic drugs), auditory hallucinations occurred more than 5 times a day for more than 6 months
5. Stable antipsychotic medication 4 weeks before and during the treatment (except auditory hallucination symptoms)

Exclusion Criteria:

1. A history of epilepsy, convulsions, stroke or other serious brain diseases
2. There are serious infectious diseases, malignant tumors, and severe somatic comorbidity
3. Mental retardation, personality disorder and so on
4. Contraindications for magnetic resonance imaging
5. Diagnose of substance dependence or abuse as primary clinical problem
6. Pregnancy
7. Participants had received Modified Electraconvulsive Therapy (MECT) or TMS treatment in recent 6 months

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Psychotic Symptom Rating Scales-Auditory Hallucination Subscale (PSYRATS-AH) | From baseline to 10 weeks
  The Psychotic Symptom Rating Scales-Auditory Hallucination Subscale (PSYRATS-AH) is an instrument designed to quantify the severity of hallucinations before and after treatment at different follow up point. Raw score range is 0-44. A higher score indicates a worse outcome.
Structural and Function MRI data | From baseline to 10 weeks
  A 3.0 T Siemens scanner was used to obtain the fMRI images in the Second Xiangya Hospital of Central South University.The MRI data wii be obtained before and after treatment at different follow up point.
Positive and Negative Syndrome Scale (PANSS) | From baseline to 10 weeks
  The PANSS total scores, subscale scores were used to evaluate the severity of psychotic symptoms for schizophrenia before and after treatment at different follow up point.The total score of the PANSS was more than 60.The higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | From baseline to 10 weeks
  Pre-post assessment of cognitive function via Repeatable Battery for the Assessment of Neuropsychological Status (RBANS)
The Stroop test | From baseline to 10 weeks
  Pre-post assessment of cognitive function via the Stroop test
Wisconsin Card Sorting Test (WCST) | From baseline to 10 weeks
  Pre-post assessment of cognitive function via Wisconsin Card Sorting Test (WCST)

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Guo, Principal Investigator — Central South University
Locations (1):
- The Second Xiangya Hospital of Central South University, Changsha, China